CLINICAL TRIAL: NCT01958333
Title: The Effects of Medium-Term Exercise Program on Health-Related Physical Fitness and Biochemical Outcomes in High-Risk Employees
Brief Title: Muscular and Metabolic Adaptations to Exercise to Benefit High-Risk Workforce
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Sergej M. Ostojic, MD, PhD, Head of Exercise Physiology Laboratory, Center for Health Sciences, Serbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-300613
Record Dates: First submitted 2013-09-29; First posted 2013-10-09 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Sedentary Lifestyle
Keywords: Health-Related Physical Fitness; Aerobic Endurance; Muscular Endurance; Flexibility
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise 1 (Experimental): Low-intensity, low-volume cardiorespiratory exercise and strength training
  Interventions: Procedure: Exercise 1
- Exercise 2 (Experimental): Medium-intensity, medium-volume cardiorespiratory exercise and strength training
  Interventions: Procedure: Exercise 2
- Exercise 3 (Experimental): High-intensity, High-volume cardiorespiratory exercise and strength training
  Interventions: Procedure: Exercise 3

INTERVENTIONS:
Procedure: Exercise 1 — Low-intensity, low-volume cardiorespiratory exercise and strength training
  Arms: Exercise 1
Procedure: Exercise 2 — Medium-intensity, Medium-volume cardiorespiratory exercise and strength training
  Arms: Exercise 2
Procedure: Exercise 3 — High-intensity, High-volume cardiorespiratory exercise and strength training
  Arms: Exercise 3

SUMMARY:
The purpose of this study is to investigate the effects of three different exercise programs (e.g. low-intensity, medium-intensity, high-intensity) administered for six months on health-related physical fitness, biochemical variables and general health outcomes in high-risk employees, with about 2000 volunteers will participate in the randomized and repeated-measure study.

DETAILED DESCRIPTION:
Exercise programs (e.g. low-intensity, medium-intensity, high-intensity) consist of aerobic workout, strength training and flexibility exercise, with different program has different intensity, volume, frequency and duration of exercise.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age

Exclusion Criteria:

* no diseases of musculoskeletal system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2114 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory endurance | Baseline and 6 months after intervention

SECONDARY OUTCOMES:
Muscular endurance | Baseline and 6 months after intervention

OTHER OUTCOMES:
Muscular strength | Baseline and 6 months after intervention
Body composition | Baseline and 6 months after intervention
Flexibility | Baseline and 6 months after intervention
AHA/ACSM risk score | Baseline and 6 months after intervention
PAR-Q score | Baseline and 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sergej M Ostojic, MD, PhD, Principal Investigator — Center for Health, Exercise and Sport Sciences
Locations (1):
- Center for Health, Exercise and Sport Sciences, Belgrade, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andres KL, Renn TA, Gray DA, Englund JM, Olsen GW, Letourneau BK. Evaluation of a cardiovascular Risk Reduction Program at a workplace medical clinic. Workplace Health Saf. 2013 Oct;61(10):459-66; quiz 467. doi: 10.1177/216507991306101006. Epub 2013 Sep 23. PMID 24053219
- [Background] Smith K. Evaluation of a stretching program to increase worker flexibility. Workplace Health Saf. 2013 Aug;61(8):329-32. doi: 10.1177/216507991306100802. PMID 23930658
- [Background] Birdee GS, Byrne DW, McGown PW, Rothman RL, Rolando LA, Holmes MC, Yarbrough MI. Relationship between physical inactivity and health characteristics among participants in an employee-wellness program. J Occup Environ Med. 2013 May;55(5):514-9. doi: 10.1097/JOM.0b013e31827f37d7. PMID 23618884